CLINICAL TRIAL: NCT06903182
Title: Preoperative TAP Block Versus Postoperative TAP Block in Patients Undergoing Laparoscopic Cholecystectomy: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Medical Doctor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6126/AO/24
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: TAP Block
Keywords: TAP block; laparoscopic cholecistectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be masked as the intervention (TAP block) will be performed after induction of general anesthesia Outcome assessor will be unaware of the group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative TAP block (Experimental): Patients will receive a preoperative TAP block with 40 mL (20 mL on the right side + 20 mL on the left side) of Ropivacaine 0.4%
  Interventions: Procedure: Preoperative TAP Block
- Postoperative TAP block (Active Comparator): Patients will receive a postoperative TAP block with 40 mL (20 mL on the right side + 20 mL on the left side) of Ropivacaine 0.4%
  Interventions: Procedure: Postoperative TAP block

INTERVENTIONS:
Procedure: Preoperative TAP Block — Patients will receive preoperative TAP block
  Arms: Preoperative TAP block
Procedure: Postoperative TAP block — Patients will receive postoperative TAP block
  Arms: Postoperative TAP block

SUMMARY:
The goal of this clinical trial is to learn if the regional anesthesia technique "TAP block" provide more analgesia when performed before or after the surgery. The main questions it aims to answer are:

Does preoperative TAP block provide greater analgesia than postoperative TAP block? Patients receiving preoperative TAP block will have less pain and take less painkillers than patients receiving postoperative TAP block?

Participants will:

Receive preoperative or postoperative TAP block They will be asked about their pain levels during the hospital stay.

DETAILED DESCRIPTION:
The TAP block is a safe, easy-to-perform, and effective technique for managing postoperative pain. It reduces opioid consumption and increases patient satisfaction. Despite recent studies indicating that postoperative TAP block might be more effective than preoperative TAP block in reducing opioid use within 24 hours, the optimal timing of its administration (before or after surgery) remains unclear.

In this study we will compare preoperative to postoperative TAP block in patients undergoing laparoscopic cholecistectomy.

The primary aim of this study is to determine the difference in postoperative pain control between preoperative and postoperative TAP block administration in patients undergoing laparoscopic cholecystectomy.

The primary objective will be to evaluate the difference in postoperative pain at rest, 24 hours after surgery, between patients receiving preoperative versus postoperative TAP block. Pain will be assessed using the Numeric Rating Scale (NRS) from 0 to 10.

Secondary objectives will be intraoperative and postoperative opioids, postoperative nausea and vomiting, pain at resnt and on movement at 0,6,12,24 hours.

ELIGIBILITY:
Inclusion Criteria

* ASA I-II patients
* Age >18 years
* Informed consent

Exclusion Criteria

* History of chronic pain
* Beta-blocker therapy
* Allergy to the drugs used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient reported pain on movement at 24 hours after the surgery | At the 24th hour after the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)

SECONDARY OUTCOMES:
Patient reported pain on movement (cough) at the end of the surgery | At the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)
Patient reported pain on rest at the end of the surgery | At the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)
Patient reported pain on rest at 6 hours after the surgery | At the 6th hour after the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)
Patient reported pain on movement at 6 hours after the surgery | At the 6th hour after the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)
Patient reported pain on rest at 12 hours after the surgery | At the 12th hour after the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)
Patient reported pain on movement at 12 hours after the surgery | At the 12th hour after the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)
Patient reported pain on rest at 24 hours after the surgery | At the 24th hour after the end of the surgery.
  Pain will be assessed with the 11 points NRS scale (0-10)
Difference in intraoperative opioids | From the enrollment to the extubation
  Difference in intraoperative fentanest in micrograms
Difference in postoperative opioids | From the extubation to the 24th postoperative hours
  Difference in postoperative morphine in milligrams
Number of participants experiencing postoperative nausea and vomiting | From extubation to the 24th postoperative hour
  Patients will be asked to report nausea and or vomiting in the postoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padua, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No